CLINICAL TRIAL: NCT02633397
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled Multi-Center Study to Assess the Safety, Tolerability, and Efficacy of Riociguat in Patients With Sickle Cell Diseases
Brief Title: A Multi-Center Study of Riociguat in Patients With Sickle Cell Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mark Gladwin (Other)
Responsible Party: Sponsor-Investigator, Mark Gladwin, Chariman of the Department of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO15110016
Record Dates: First submitted 2015-12-07; First posted 2015-12-17 (Estimated); Results first posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Sickle Cell Disease
Keywords: SCD; Sickle Cell Disease; Riociguat; Adempas
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Riociguat (Experimental): Treatment Arm
  Interventions: Drug: Riociguat
- Placebo (Placebo Comparator): Placebo Arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riociguat — Riociguat 0.5 mg, 1.0 mg, 1.5 mg, 2.0 mg and 2.5 mg three times a day for 12 weeks
  Other Names: Adempas
  Arms: Riociguat
Drug: Placebo — Matching placebo to riociguat 0.5 mg, 1.0 mg, 1.5 mg, 2.0 mg and 2.5 mg three times a day for 12 weeks
  Arms: Placebo

SUMMARY:
The proposed study is a Phase 2 multi-center, randomized, double-blind, placebo-controlled, parallel groups study aimed to evaluate the safety, tolerability and the efficacy of riociguat compared with placebo in patients with sickle cell disease (SCD).

DETAILED DESCRIPTION:
This randomized study involves 12 weeks of treatment with riociguat pills or placebo pills, and a follow-up period of 30 days after treatment. The dose is adjusted every 2 weeks based on systolic blood pressure (SBP) and well-being assessed at that visit. Physical examinations, vital signs, blood tests and questionnaires will be performed at 2 week intervals during the double blinded study treatment. Echocardiogram, urine testing, six-minute walk distance and questionnaires will be assessed at the beginning and end of the treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Sickling disorder (HbSS, HbSC, HbSbeta-thalassemia, HbSD, HbSO-Arab documented by hemoglobin electrophoresis or HPLC fractionation)
* At least one of the following findings: a. Systolic blood pressure ≥ 130 mm Hg on at least two occasions at least 1 day apart (one of these may be by history), b. Macroalbuminuria as manifested by urine albumin to creatinine ratio > 300 mg/g, c. Tricuspid regurgitant velocity (TRV) > 2.9 m/sec measured by echocardiography d. NT-proBNP level ≥ 160 pg/mL e. Urinalysis protein 1 + or higher.
* Females of reproductive potential (FRP) must have a negative, pre-treatment pregnancy test. Post-menopausal women (defined as no menses for at least 1 year or post-surgical from bilateral oophorectomy) are not required to undergo a pregnancy test.
* Females of reproductive potential must agree to use reliable contraception when sexually active. Adequate contraception is defined as any combination of at least 2 effective methods of birth control, of which at least one is a physical barrier (e.g. condoms with hormonal contraception or implants or combined oral contraceptives, certain intrauterine devices). Adequate contraception is required beginning at the signing of the informed consent form until one month after the last dose of riociguat.
* Patients must be willing to provide a blood sample for DNA analysis.

Exclusion Criteria:

* Pregnant or breast feeding women
* Patients with severe hepatic impairment defined as Child Pugh C
* End stage renal disease requiring dialysis
* Patients with eGFR <30 mL/min/1.73m, where GFR is estimated based on CKD-epi equation
* Patients on phosphodiesterase type 5 inhibitors (PDE-5) (such as sildenafil, tadalafil, vardenafil) and nonspecific PDE inhibitors (such as dipyridamole or theophylline) or nitrates
* Patients on strong cytochrome P450 (CYP) and P-glycoprotein 1(P-gp)/BCRP inhibitors such as systemic azole antimycotics (eg: ketoconazole, itraconazole), or HIV protease inhibitors (such as ritonavir)
* Patients on St. John's Wort
* If patients are taking antihypertensive drugs, hydroxyurea, L-glutamine, crizanlizumab, or voxelotor prior to enrollment, they are excluded until the dose level is stable for at least three months
* Systolic blood pressure <95 mm Hg at Screening Visit 1 or 2 or Week 0 before randomization
* Current enrollment in an investigational new drug trial. Patients are eligible for enrollment 30 days after the last dose of an investigational drug has been received
* Evidence of qualitative urine drug test at screening for cocaine, phencyclidine (PCP), heroin, or amphetamines within three months prior to enrollment
* Patients who have recently (last six months) experienced serious bleeding from the lung or have undergone a bronchial arterial embolization procedure.
* Pulmonary hypertension associated with Idiopathic Interstitial Pneumonias
* Medical disorder, condition, or history that in the investigator's judgment would impair the patient's ability to participate or complete this study or render the patient to be inappropriate for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gladwin, MD, Principal Investigator — University of Pittsburgh
Locations (20):
- United States (20):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Howard University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Illinois, Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Tulane University, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - New York Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Albert Einstein University/ Montefiore Medical Center, The Bronx, New York
  - UNC Comprehensive Sickle Cell Center, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Ohio State University, Columbus, Ohio
  - UPMC Division of Hematology and Oncology, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Virginia Commonwealth University Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gladwin MT, Gordeuk VR, Desai PC, Minniti C, Novelli EM, Morris CR, Ataga KI, De Castro L, Curtis SA, El Rassi F, Ford HJ, Harrington T, Klings ES, Lanzkron S, Liles D, Little J, Nero A, Smith W, Taylor JG 6th, Baptiste A, Hagar W, Kanter J, Kinzie A, Martin T, Rafique A, Telen MJ, Lalama CM, Kato GJ, Abebe KZ. Riociguat in patients with sickle cell disease and hypertension or proteinuria (STERIO-SCD): a randomised, double-blind, placebo controlled, phase 1-2 trial. Lancet Haematol. 2024 May;11(5):e345-e357. doi: 10.1016/S2352-3026(24)00045-0. Epub 2024 Mar 27. PMID 38554715
- [Derived] Azbell RCG, Desai PC. Treatment dilemmas: strategies for priapism, chronic leg ulcer disease, and pulmonary hypertension in sickle cell disease. Hematology Am Soc Hematol Educ Program. 2021 Dec 10;2021(1):411-417. doi: 10.1182/hematology.2021000275. PMID 34889382

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Riociguat | Placebo
Started | 66 | 64
Completed | 50 | 47
Not Completed | 16 | 17
Not completed — Adverse Event | 8 | 8
Not completed — Study Burden | 4 | 1
Not completed — Treatment interruption | 2 | 5
Not completed — Death | 2 | 2
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riociguat | Placebo | Total
Number analyzed (Participants) | 66 | 64 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at screening
  years | 41.0 (11.8) | 44.8 (12.3) | 42.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 30 | 28 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 63 | 61 | 124
  Unknown or Not Reported | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 63 | 64 | 127
  Race: Some Other Race | 2 | 0 | 2
  Race: Unknown | 1 | 0 | 1
Clinical Sickle Cell Phenotype (as reported by site) [Count of Participants; unit: Participants]
  SCD, subtype not immediately available | 0 | 1 | 1
  HbSS | 49 | 48 | 97
  HbSC | 13 | 11 | 24
  HbSbeta-zero-thalassemia | 3 | 1 | 4
  HbSbeta-plus-thalassemia | 1 | 3 | 4
BMI [Mean (Standard Deviation); unit: kg/m²] — Body Mass Index Population: Four participants had a missing result
  kg/m²
    number analyzed (Participants) | 64 | 62 | 126
    (all) | 29.2 (9.7) | 27.0 (6.2) | 28.1 (8.2)
Systolic BP [Mean (Standard Deviation); unit: mmHg] | 128.5 (17.8) | 125.5 (15.6) | 127.1 (16.7)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 76.7 (11.5) | 73.8 (11.2) | 75.3 (11.4)
Stage 1 hypertension [Count of Participants; unit: Participants] — Systolic BP ≥130 or diastolic BP ≥80
  Participants
    No | 30 | 28 | 58
    Yes | 36 | 36 | 72
Heart rate [Mean (Standard Deviation); unit: beats per minute] | 84.4 (12.4) | 81.2 (13.9) | 82.8 (13.2)
Mean arterial pressure (MAP) [Mean (Standard Deviation); unit: mmHg] | 94.0 (12.4) | 91.1 (11.1) | 92.5 (11.8)
Pain severity score [Mean (Standard Deviation); unit: Score on a scale] — Assessed by the Brief Pain Inventory (BPI) Short Form - score ranges from 0 (no pain) to 10 (Pain as bad as you can imagine).
  Score on a scale | 3.5 (2.2) | 3.2 (2.5) | 3.4 (2.4)
Pain interference score [Mean (Standard Deviation); unit: Score on a scale] — Assessed by the Brief Pain Inventory (BPI) short form - score ranges from 0 (does not interfere) to 10 (completely interferes).
  Score on a scale | 3.1 (2.7) | 3.0 (2.8) | 3.1 (2.8)
6-Minute Walk Test (6MWT) [Mean (Standard Deviation); unit: meters] — The distance walked in six minutes was used to assess the exercise capacity of the patient at baseline Population: three participants are missing results.
  meters
    number analyzed (Participants) | 64 | 63 | 127
    (all) | 416.9 (154.0) | 374.0 (127.9) | 395.6 (142.7)
6-Minute Walk Test (6MWT) [Count of Participants; unit: Participants] — The distance walked in six minutes was used to assess the exercise capacity of the patient at baseline. Population: three participants are missing results.
  Participants
    <333 meters: number analyzed (Participants) | 64 | 63 | 127
    <333 meters | 17 | 18 | 35
    ≥333 - ≤450 meters: number analyzed (Participants) | 64 | 63 | 127
    ≥333 - ≤450 meters | 31 | 35 | 66
    >450 meters: number analyzed (Participants) | 64 | 63 | 127
    >450 meters | 16 | 10 | 26
TR velocity [Mean (Standard Deviation); unit: peak, m/s] | 2.37 (0.61) | 2.45 (0.70) | 2.41 (0.66)
TR velocity [Count of Participants; unit: Participants]
  <2.5 m/s | 37 | 35 | 72
  ≥2.5 - <3 m/s | 22 | 15 | 37
  ≥3 m/s | 7 | 14 | 21
Ejection fraction [Mean (Standard Deviation); unit: Percentage] — Biplane measurement Population: Two participants are missing results.
  Percentage
    number analyzed (Participants) | 65 | 63 | 128
    (all) | 59.42 (5.95) | 60.86 (6.28) | 60.13 (6.13)
Macroalbuminuria [Count of Participants; unit: Participants] — Urine albumin to creatinine ratio >300 mg/g at screening. Screening labs for macroalbuminuria were up to 12 months before enrollment.
  Participants
    No | 46 | 39 | 85
    Yes | 20 | 25 | 45
Albumin/Creatinine Ratio (ACR) [Mean (Standard Deviation); unit: mg/g] — Population: Unavailable data for Twenty participants. ACR was undetectable in 11 participants, while 9 participants had missing data.
  mg/g
    number analyzed (Participants) | 55 | 55 | 110
    (all) | 249.1 (379.4) | 361.7 (849.5) | 305.4 (657.3)
Albuminuria [Count of Participants; unit: Participants] — Population: Unavailable data for Twenty participants. ACR was undetectable in 11 participants, while 9 participants had missing data.
  Participants
    number analyzed (Participants) | 55 | 55 | 110
    Normal (ACR<30mg/g) | 18 | 14 | 32
    Microalbuminuria (ACR 30-300mg/g) | 25 | 28 | 53
    Macroalbuminuria (ACR >300mg/g) | 12 | 13 | 25
GFR [Mean (Standard Deviation); unit: ml/min/1.73 m²] | 114.5 (28.0) | 105.4 (34.3) | 110.0 (31.5)
Ever smoked cigarettes [Count of Participants; unit: Participants]
  No | 47 | 49 | 96
  Yes | 19 | 15 | 34
Ever had a blood transfusion [Count of Participants; unit: Participants]
  No | 7 | 2 | 9
  Yes | 59 | 62 | 121

OUTCOME MEASURES:

1. Primary Outcome: Overall Incidence of Treatment Emergent Severe Adverse Events (SAE)
Description: The primary endpoint was the proportion of participants who experienced at least 1 treatment-emergent serious adverse event (SAE), which was defined as any event occurring after the baseline visit (i.e., after initiation of study drug), adjudicated by a designated committee of protocol investigators and outside experts. SAEs were considered to be treatment-emergent if they started or worsened after the first dose of study medication and up to 7 days after end of study treatment.
Time Frame: Baseline through 7 days after discontinuation of treatment, up to 13 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
Participants | 15 | 20
Statistical Analysis 1: Comparison: Riociguat vs Placebo; P- Value was the exact logistic regression adjusted for clinical site; Test type: Superiority; p = 0.19, Regression, Logistic

2. Secondary Outcome: Frequency of SAE Due to Sickle Cell Related Painful Crisis
Description: The proportion of participants with treatment-emergent SAE for sickle-cell related crises (Vaso-occlusive crises)
Time Frame: Baseline through 7 days after discontinuation of treatment, up to 13 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
Participants | 11 | 14
Statistical Analysis 1: Comparison: Riociguat vs Placebo; P- Value was the exact logistic regression adjusted for clinical site; Test type: Superiority; p = 0.42, Regression, Logistic

3. Secondary Outcome: Overall Incidences of Treatment-emergent Adverse Events (AEs)
Description: Proportion of participants that experienced treatment-emergent AEs
Time Frame: Baseline to Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
Participants | 53 | 45
Statistical Analysis 1: Comparison: Riociguat vs Placebo; P- Value was the exact logistic regression adjusted for clinical site; Test type: Superiority; p = 0.52, Regression, Logistic

4. Secondary Outcome: Incidences of Sickle Cell Related Clinical Complications
Description: Incidence of Vaso-occlusive Crisis (VOC) between baseline and week 12
Time Frame: Baseline to Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
Participants | 23 | 21

5. Secondary Outcome: Pain Intensity Using the Brief Pain Inventory
Description: Brief Pain Inventory (BPI) short form - score ranges from 0 (no pain) to 10 (Pain as bad as you can imagine)
  Mean at 12 weeks assessed using ANCOVA adjusting for baseline.
Time Frame: Baseline, 12 weeks
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
score on a scale | 3.18 [2.75 to 3.62] | 3.32 [2.88 to 3.75]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; ANCOVA model adjusted for clinic site; Test type: Superiority; p = 0.69, ANCOVA; Mean Difference (Final Values) = -0.14, 90% CI 2-sided [-0.70 to 0.42]

6. Secondary Outcome: 6-minute Walk Distance
Description: 6-minute walk distance was used to assess functional exercise capacity
  Mean at 12 weeks assessed using ANCOVA adjusting for baseline.
Time Frame: Baseline, 12 weeks
Measure: Mean (90% Confidence Interval); unit: meters
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
meters | 391.97 [332.29 to 451.66] | 431.49 [369.61 to 493.37]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; ANCOVA model adjusted for clinic site; Test type: Superiority; p = 0.40, ANCOVA; Mean Difference (Final Values) = -39.51, 90% CI 2-sided [-117.05 to 38.02]

7. Secondary Outcome: Changes in the Dyspnea Borg Scale
Description: Baseline to 12 weeks mean change of the Borg dyspnea scores, post 6MWT, using a linear regression model.
  Dyspnea Borg score was used to measure the level of severity of breathlessness perceived by the patient at the end of the 6MWD Test. The severity is measured on a 10-point scale with 0= nothing at all and 10=maximum severity of breathlessness.
Time Frame: Baseline,12 Weeks
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
score on a scale | 0.50 [0.17 to 0.83] | 0.20 [-0.14 to 0.53]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; Linear regression model adjusted for clinic site; Test type: Superiority; p = 0.23, Regression, Linear; Mean Difference (Final Values) = 0.31, 90% CI 2-sided [-0.11 to 0.73]

8. Secondary Outcome: Fatigue Borg Scale
Description: Fatigue Borg score was used to rank the participant's exertion at the end of the 6MWD Test. The rate of exertion was given according to a scale ranging from 0 (nothing at all) to 10=maximum severity of exertion
  Mean at 12 weeks assessed using ANCOVA adjusting for baseline.
Time Frame: Baseline,12 weeks
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
score on a scale | 1.95 [1.53 to 2.37] | 2.03 [1.6 to 2.46]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; ANCOVA model adjusted for clinic site; Test type: Superiority; p = -0.80, ANCOVA; Mean Difference (Final Values) = -0.08, 90% CI 2-sided [-0.62 to 0.46]

9. Secondary Outcome: Changes in Blood Pressure as the Main Pharmacodynamic (MAP)
Description: Baseline to 12 weeks mean change of MAP, estimated with a repeated measures analysis (Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks) using a linear mixed model.
Time Frame: Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks
Measure: Mean (90% Confidence Interval); unit: mmHg
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
mmHg | -8.20 [-10.48 to -5.91] | -1.24 [-3.58 to 1.10]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; Linear mixed model with random intercept was used to compare the change in MAP as a function of time, the interaction between time and study arm, and clinic site; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -6.96, 90% CI 2-sided [-10.22 to -3.69]

10. Secondary Outcome: Tricuspid Regurgitant Velocity (TRV) Using Non-invasive Echocardiography
Description: Mean TRV at 12 weeks assessed using ANCOVA, adjusting for baseline.
Time Frame: Baseline, 12 Weeks
Measure: Mean (90% Confidence Interval); unit: m/s
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
m/s | 2.17 [2.04 to 2.30] | 2.31 [2.19 to 2.44]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; ANCOVA model adjusted for clinic site; Test type: Superiority; p = 0.15, ANCOVA; Mean Difference (Final Values) = -0.14, 90% CI 2-sided [-0.31 to 0.02]

11. Secondary Outcome: End-systolic Volume Using Non-invasive Echocardiography
Description: Mean end-systolic volume (biplane) at 12 weeks, assessed using ANCOVA adjusting for baseline.
Time Frame: Baseline,12 weeks
Measure: Mean (90% Confidence Interval); unit: ml
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
ml | 46.40 [43.59 to 49.22] | 53.1 [50.33 to 55.88]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; ANCOVA model adjusted for clinic site; Test type: Superiority; p = 0.003, ANCOVA; Mean Difference (Final Values) = -6.70, 90% CI 2-sided [-10.28 to -3.12]

12. Secondary Outcome: Ejection Fraction (Biplane) Using Non-invasive Echocardiography
Description: Mean ejection fraction (biplane) at 12 weeks, assessed using ANCOVA adjusting for baseline.
Time Frame: Baseline, 12 weeks
Measure: Mean (90% Confidence Interval); unit: percentage
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
percentage | 63.19 [62.01 to 64.37] | 59.67 [58.51 to 60.83]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; ANCOVA model adjusted for clinic site; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.52, 90% CI 2-sided [2.00 to 5.04]

13. Secondary Outcome: Changes in the Levels of Plasma NT-proBNP
Description: Mean Change in the levels of plasma NT-proBNP from baseline to 12 weeks using a linear regression model.
Time Frame: Baseline,12 weeks
Measure: Mean (90% Confidence Interval); unit: pg/mL
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
pg/mL | 54.67 [-477.91 to 587.2] | -231.89 [-780.36 to 316.5]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; Linear regression model adjusted for clinic site; Test type: Superiority; p = 0.51, Regression, Linear; Mean Difference (Final Values) = 286.56, 90% CI 2-sided [-429.86 to 1002.99]

14. Secondary Outcome: Changes in Albumin/Creatinine Ratio
Description: Albumin/Creatinine Ratio (ACR) mean change from baseline to 12 weeks using linear regression model.
Time Frame: Baseline,12 weeks
Measure: Mean (90% Confidence Interval); unit: mg/g
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
mg/g | -56.96 [-126.10 to 12.17] | 25.22 [-44.66 to 95.11]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; Linear regression model adjusted for clinic site; Test type: Superiority; p = 0.14, Regression, Linear; Mean Difference (Final Values) = -82.18, 90% CI 2-sided [-173.69 to 9.32]

15. Secondary Outcome: Microalbuminuria
Description: Odds ratio per week of microalbuminuria estimated with a repeated measures analysis (baseline, 12 weeks) using a generalized linear mixed model without random slope
Time Frame: Baseline,12 weeks
Population: Participants with undetectable ACR or macroalbuminuria (>300 ACR) were excluded
Measure: Number (90% Confidence Interval); unit: odds ratio
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 43 | 42
odds ratio | 0.96 [0.87 to 1.06] | 0.94 [0.85 to 1.04]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; Generalized linear mixed model (logit link) with random intercept was used to compare microalbuminuria frequency as a function of time and the interaction between time and study arm; Test type: Superiority; p = 0.78, Mixed Models Analysis

16. Secondary Outcome: Macroalbuminuria
Description: Odds ratio per week of macroalbuminuria estimated with a repeated measures analysis (baseline, 12 weeks) using a generalized linear mixed model without random slope.
Time Frame: Baseline,12 weeks
Population: Participants with undetectable ACR or microalbuminuria (30-300 ACR) were excluded
Measure: Number (90% Confidence Interval); unit: odds ratio
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 30 | 27
odds ratio | 1.03 [0.81 to 1.31] | 0.84 [0.66 to 1.08]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; Generalized linear mixed model (logit link) with random intercept was used to compare macroalbuminuria frequency as a function of time and the interaction between time and study arm; Test type: Superiority; p = 0.30, Mixed Models Analysis

17. Secondary Outcome: Changes in Glomerular Filtration Rate
Description: Mean change in GFR to 12 weeks, estimated with a repeated measures analysis (Baseline, 4 weeks, 8 weeks, 12 weeks) a using a linear mixed model.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Measure: Mean (90% Confidence Interval); unit: ml/min/1.73 m²
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
ml/min/1.73 m² | -4.13 [-7.11 to -1.14] | 0.79 [-2.29 to 3.87]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; Linear mixed model with random intercept was used to compare the change in GFR as a function of time, the interaction between time and study arm, and clinic site; Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = -4.91, 90% CI 2-sided [-9.21 to -0.62]

18. Secondary Outcome: Chronic Kidney Disease (CKD) Stage - Low Risk Versus at Least Moderately Increased Risk
Description: Odds ratio (OR) per week of low-risk CKD stage versus at least moderately increased risk (includes moderately increased risk CKD, high increased risk CKD, and very high increased risk CKD) estimated with a repeated measures analysis (baseline, 12 weeks) using a generalized linear mixed model without random slope
Time Frame: Baseline,12 weeks
Measure: Number (90% Confidence Interval); unit: odds ratio
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
odds ratio | 0.99 [0.90 to 1.08] | 0.95 [0.86 to 1.04]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; Generalized linear mixed model (logit link) with random intercept was used to compare CKD stage frequency as a function of time and the interaction between time and study arm; Test type: Superiority; p = 0.56, Mixed Models Analysis

19. Secondary Outcome: Changes in Hemoglobin
Description: Mean change in hemoglobin to 12 weeks, estimated with a repeated measures analysis (Baseline, 4 weeks, 8 weeks, 12 weeks) a using a linear mixed model.
Time Frame: Baseline, 4 weeks, 8 weeks,12 weeks
Measure: Mean (90% Confidence Interval); unit: g/dL
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
g/dL | -0.21 [-0.40 to -0.01] | 0.04 [-0.16 to 0.24]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; Linear mixed model with random intercept was used to compare the change in hemoglobin as a function of time, the interaction between time and study arm, and clinic site; Test type: Superiority; p = 0.15, Mixed Models Analysis; Mean Difference (Final Values) = -0.24, 90% CI 2-sided [-0.52 to 0.03]

20. Secondary Outcome: Changes in Reticulocyte Count
Description: Mean change in reticulocyte count to 12 weeks, estimated with a repeated measures analysis (Baseline, 4 weeks, 8 weeks, 12 weeks) a using a linear mixed model.
Time Frame: Baseline, 4 weeks, 8 weeks,12 weeks
Measure: Mean (90% Confidence Interval); unit: percentage
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
percentage | 0.32 [-0.54 to 1.19] | -1.15 [-2.05 to -0.24]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; Linear mixed model with random intercept was used to compare the change in reticulocyte count as a function of time, the interaction between time and study arm, and clinic site; Test type: Superiority; p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 1.47, 90% CI 2-sided [0.22 to 2.72]

21. Secondary Outcome: Changes in White Blood Cell Count
Description: Mean change in White Blood Cell count to 12 weeks estimated with a repeated measures analysis (Baseline, 4 weeks, 8 weeks, 12 weeks) a using a linear mixed model.
Time Frame: Baseline, 4 weeks, 8 weeks,12 weeks
Measure: Mean (90% Confidence Interval); unit: (x10^9 cells/L)
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
(x10^9 cells/L) | -0.28 [-0.83 to 0.26] | -0.13 [-0.69 to 0.43]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; Linear mixed model with random intercept was used to compare the change in WBC count as a function of time, the interaction between time and study arm, and clinic site; Test type: Superiority; p = 0.75, Mixed Models Analysis; Mean Difference (Final Values) = -0.15, 90% CI 2-sided [-0.93 to 0.63]

22. Secondary Outcome: Changes in Lactate Dehydrogenase (LDH)
Description: Mean change in LDH to 12 weeks estimated with a repeated measures analysis (Baseline, 4 weeks, 8 weeks, 12 weeks) a using a linear mixed model.
Time Frame: Baseline, 4 weeks, 8 weeks,12 weeks
Measure: Mean (90% Confidence Interval); unit: U/L
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
U/L | -43.30 [-67.49 to -19.10] | -14.02 [-39.80 to 11.76]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.17, Mixed Models Analysis; Mean Difference (Final Values) = -29.28, 90% CI 2-sided [-64.63 to 6.08]

23. Secondary Outcome: Changes in Fetal Hemoglobin
Description: Mean change in fetal hemoglobin from baseline to 12 weeks using a linear mixed model
Time Frame: Baseline,12 weeks
Measure: Mean (90% Confidence Interval); unit: Percentage
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 66 | 64
Percentage | -1.91 [-3.05 to -0.78] | -0.28 [-1.44 to 0.88]
Statistical Analysis 1: Comparison: Riociguat vs Placebo; Linear regression model adjusted for clinic site; Test type: Superiority; p = 0.07, Regression, Linear; Mean Difference (Final Values) = -1.64, 90% CI 2-sided [-3.13 to -0.15]

ADVERSE EVENTS:
Time Frame: Adverse events were data collected from baseline through 7 days after discontinuation of treatment, up to 13 Weeks
Description: Adverse events and deaths were not collected by dose level.
Arm/Group | Riociguat | Placebo
All-Cause Mortality (participants affected / at risk) | 2/66 | 2/64
Serious Adverse Events (participants affected / at risk) | 15/66 | 20/64
Other Adverse Events (participants affected / at risk) | 53/66 | 45/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat (N=66) | Placebo (N=64)
VOC (General disorders) | 11 (17) | 14 (23)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Mitral Valve Disease (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Other - Pyelonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Other - Dizziness (Endocrine disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Other - Papilledema (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat (N=66) | Placebo (N=64)
VOC (General disorders) | 23 (65) | 21 (46)
Malaise (General disorders) | 3 (3) | 3 (3)
Fatigue (General disorders) | 3 (3) | 2 (2)
Edema Limbs (General disorders) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 9 (11) | 8 (9)
Nausea (Gastrointestinal disorders) | 7 (8) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 4 (5) | 4 (5)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 8 (8) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Other (Gastrointestinal disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 14 (16) | 6 (7)
Dizziness (Nervous system disorders) | 8 (9) | 3 (4)
Other (Musculoskeletal and connective tissue disorders) | 9 (15) | 10 (14)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Palpitations (Cardiac disorders) | 5 (5) | 2 (2)
Chest Pain - Cardiac (Cardiac disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT02633397/Prot_SAP_000.pdf